CLINICAL TRIAL: NCT04243044
Title: Neuromodulation of Spinal Circuits: Effects on Spasticity, Nociception, and Motor Activation
Brief Title: Influence of Transcutaneous Spinal Stimulation Intensity on Spasticity After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Edelle Field-Fote, PT, PhD, Director, Spinal Injury Research & The Hulse Spinal Injury Laboratory, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1343378
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Intensity 1 (0.8x reflex threshold, continuous, 30 minute duration) (Experimental): Transcutaneous spinal stimulation will be applied continuously at 0.8x reflex threshold as determined from baseline testing of posterior root muscle reflexes.
  Interventions: Device: Transcutaneous spinal stimulation
- Intensity 2 (0.8x reflex threshold, dual-site, 30 minute duration) (Experimental): Transcutaneous spinal stimulation will be applied continuously at two sites at 0.8x reflex threshold as determined from baseline testing of posterior root muscle reflexes.
  Interventions: Device: Transcutaneous spinal stimulation
- Intensity 3 (0.8x reflex threshold, burst, 30 minute duration) (Experimental): Transcutaneous spinal stimulation will be applied in bursts at 0.8x reflex threshold as determined from baseline testing of posterior root muscle reflexes.
  Interventions: Device: Transcutaneous spinal stimulation

INTERVENTIONS:
Device: Transcutaneous spinal stimulation — Transcutaneous spinal stimulation will be delivered for 30 minutes using biphasic stimulation with a single round electrode as the cathode placed directly over the spine at the T11/T12 (and the lumbar spine for dual-site stimulation) spinous interspace, and two interconnected dispersive (reference) electrodes placed on the abdomen, lateral to the umbilicus. Stimulation intensity will be set to the specified level determined through a pre-stimulation assessment (0.8x reflex threshold). Treatments will be a minimum of 48 hours apart.

SUMMARY:
Transcutaneous spinal stimulation (TSS) is a form of electrical stimulation delivered over the skin of the spine that may be valuable for reducing spasticity without the side effects of antispasticity medications. The intensity of stimulation, or dose, that promotes the best response is not known. Understanding the response to different intensities of stimulation and how they affect spasticity will help guide rehabilitation for persons with SCI. Therefore, this study aims to identify the effects of TSS as a non-drug intervention for spasticity management.

DETAILED DESCRIPTION:
Spasticity involves involuntary muscle activity in persons with spinal cord injury (SCI) that can include increased response to muscle stretch and physical touch, as well as muscle stiffness. Due to the combination of symptoms, several drug therapies are currently prescribed to reduce spasticity but they may have negative side effects including fatigue and muscle weakness. Transcutaneous spinal stimulation (TSS) is a form of electrical stimulation delivered over the skin of the spine that seems to have effects that are similar to drug therapy. Prior studies of TSS in persons with SCI suggest that TSS can reduce spasticity without negative side effects. The intensity of stimulation, or dose, that promotes the best response is not known. In addition, sensitive measurements are necessary to assess the changes that can be seen in multiple presentations of spasticity. Understanding the response to different intensities of stimulation and how they affect spasticity will help guide rehabilitation for persons with SCI. Therefore, this study aims to identify the effects of TSS as a non-drug intervention for spasticity management.

ELIGIBILITY:
Inclusion Criteria:

The participant must meet all of the following criteria to be eligible for the study:

* Ability and willingness to authorize the use of protected health information (PHI)
* Be 16 years of age or older
* Have a SCI with any severity classification (AIS A, B, C, or D) that occurred at least 3 months ago
* Have at least mild "spasticity" affecting lower extremity muscles, as indicated by a pendulum test first swing excursion angle of ≤ 77° or ≥ 5 beats of clonus on the ankle drop test
* Use of prescription medications is acceptable, as long as the dosage has not changed in the last 2 weeks and notification of medication changes is made during study participation
* Ability to follow multiple commands
* Ability to communicate pain or discomfort

Exclusion Criteria:

The presence of any one of the following criteria leads to exclusion:

* Progressive or potentially progressive spinal lesions, including degenerative, or progressive vascular disorders of the spine and/or spinal cord
* Neurologic level below spinal level T12
* History of cardiovascular irregularities (e.g. atrial fibrillation)
* Active cancer or a history of cancer
* Orthopedic pathology that would limit participation in the protocol (e.g. knee or hip flexion contractures of greater than 10 degrees)
* Use of semi-permanent or permanent anti-spasmodic treatment (i.e. botox, selective dorsal rhizotomy)
* Women who are pregnant, or who have reason to believe they are, or may become pregnant due to unknown risks to the fetus associated with TSS
* Persons who have implanted stimulators of any type will be excluded due to unknown potential of electrical stimulation effects (e.g. baclofen pump, epidural spinal stimulator, implanted cardiac defibrillator, diaphragmatic pacemaker)
* Active infection of any type, as infection may exacerbate spasticity resulting in inability to identify the influence of the treatment
* Skin irregularities, sensitivity, or lesions that would increase the risk of stimulation-associated adverse events

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Pendulum Test | Before and Immediately after each intervention session through study completion, an average of 2 weeks
  The pendulum test will be performed during which the participant will be positioned supine on a mat with the lower leg hanging over the mat. A member of the study staff will support the participant's extended lower leg and then release the leg allowing it to swing freely. Muscle activity during each maneuver will be recorded using electromyography (EMG) of the quadriceps, hamstrings, tibialis anterior, and soleus muscles of the lower extremity identified as having the greatest spasticity. Biomechanical measurements will be captured through the use of an electrogoniometer placed at the knee joint.

SECONDARY OUTCOMES:
Change in Ankle Clonus Test | Before and Immediately after each intervention session through study completion, an average of 2 weeks
  The ankle clonus test will be performed during which the participant will be seated at the edge of a mat with the lower leg hanging over the mat. A member of the study staff will support the participant's leg above a box and then release the leg allowing the front of the foot to land on the edge of the box. Muscle activity during each maneuver will be recorded using EMG of the tibialis anterior and soleus muscles of the lower extremity identified as having the greatest spasticity. Biomechanical measurements will be captured through the use of an electrogoniometer placed at the ankle joint.
Change in posterior root muscle reflexes (PRMRs) | Before and Immediately after each intervention session through study completion, an average of 2 weeks
  PRMRs will be assessed to identify the spinal stimulation threshold at which muscle activity occurs in the soleus (reflex threshold). Electrode placement as outlined for intervention will be followed for this assessment. Briefly, stimulating pulses of 1ms duration (applied via a Digitimer DS7A constant current stimulator) will be delivered through the stimulating electrodes and intensity will be gradually increased until a motor event is electrophysiologically observed in the soleus. This reflex threshold stimulation intensity will be utilized to set the parameters of the three tcSCS intervention sessions - 80% of reflex threshold (0.8xRT).
Change in Plantar Flexor Reflex Response | Before and Immediately after each intervention session through study completion, an average of 2 weeks
  Muscle activity induced through noxious sensory input will be assessed through instrumented flexor reflex response. Flexor reflex response will be tested at 1.2x reflex threshold of the tibialis anterior for three stimulus trains. Then, the noxious sensory stimulus will be standardized through electrocutaneous stimulation to the plantar surface of the participant's foot (parameters: 25mA, 500Hz, 20ms train). Muscle activity after each stimulus will be recorded using electromyography (EMG) of the quadriceps, hamstrings, tibialis anterior, and soleus muscles of the lower extremity identified as having the greatest spasticity.
Stimulation Tolerability Questionnaire | Immediately following each intervention session through study completion, an average of 2 weeks.
  Participants will be asked to rate how tolerable stimulation was during the session and to describe specific sensations that contributed to this rating.
Qualities of Spasticity Survey | Before and Immediately after each intervention session through study completion, an average of 2 weeks
  The Qualities of Spasticity Survey is a self-report questionnaire that asks participants about the physical qualities of their spasticity and how it impacts daily life. Participants will be asked to report their experience with their spasticity over the past 48 hours.
Modified Penn Spasm Frequency Scale | Before and four hours after each intervention session through study completion, an average of 2 weeks
  The Modified Penn Spasm Frequency Scale is a self-report questionnaire which asks participants to rate the frequency and severity of their spasms during the last hour.

OTHER OUTCOMES:
Modified SCI-SET | Completed during the enrollment session only.
  The Modified SCI-SET is a self-report questionnaire that asks participants to rate how their spasticity has impacted various aspects of their life over the past seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thatcher KL, Nielsen KE, Sandler EB, Daliet OJ 4th, Iddings JA, Field-Fote EC. Optimizing transcutaneous spinal stimulation: excitability of evoked spinal reflexes is dependent on electrode montage. J Neuroeng Rehabil. 2025 Jan 6;22(1):2. doi: 10.1186/s12984-024-01524-5. PMID 39762915